CLINICAL TRIAL: NCT03468907
Title: The Safety of Anti-viral Therapy in Preventing Mother-to-child Transmission of Hepatitis B Virus in Pregnant Women After Discontinuation
Brief Title: The Safety of Anti-viral Therapy in Preventing HBV MTCT in Pregnant Women After Discontinuation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chao-Shuang Lin, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Safety of anti-viral agents
Record Dates: First submitted 2018-01-21; First posted 2018-03-19 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis B, Chronic
Keywords: hepatitis B virus; exacerbation; antiviral agents; pregnancy; flare
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Telbivudine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Pregnant mothers who opt for antiviral therapy will start on oral LDT 600 mg or TDF 300 mg (as per patients' wishes) daily between gestational weeks 24 and 28. Antiviral therapy will be discontinued in intrapartum or at postpartum 6 weeks.
Masking Description: The care provider, participant, investigator and outcomes assessor all konw the process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early cessation (Experimental): Pregnant mothers who opted for antiviral therapy would start on oral LDT 600 mg or TDF 300 mg (as per patients' wishes) daily between gestational weeks 24 and 28. Antiviral therapy was discontinued in intrapartum.
  Interventions: Drug: Telbivudine 600mg; Drug: Tenofovir disoproxil fumarate 300mg
- Late cessation (Experimental): Pregnant mothers who opted for antiviral therapy would start on oral LDT 600 mg or TDF 300 mg (as per patients' wishes) daily between gestational weeks 24 and 28. After delivery, mothers ceased antiviral treatment at postpartum 6 weeks.
  Interventions: Drug: Telbivudine 600mg; Drug: Tenofovir disoproxil fumarate 300mg
- Control (No Intervention): Eligible patients who refused antiviral therapy but consented to the study were assigned to the control arm.

INTERVENTIONS:
Drug: Telbivudine 600mg — Pregnant mothers who opted for antiviral therapy would start on oral LDT 600 mg daily between gestational weeks 24 and 28.
  Other Names: Sebivo
  Arms: Early cessation; Late cessation
Drug: Tenofovir disoproxil fumarate 300mg — Pregnant mothers who opted for antiviral therapy would start on oral TDF 300 mg daily between gestational weeks 24 and 28.
  Other Names: Viread
  Arms: Early cessation; Late cessation

SUMMARY:
Mother-to-child transmission (MTCT) is the most common mode of perpetuating chronic hepatitis B virus (HBV) infection in endemic countries. Many studies have demonstrated antepartum anti-viral therapy (AVT) is a advisable option to reduce mother-to-child transmission and the risk of vaccination breakthrough in infants who received passive-active immunoprophylaxis. However, several controversies over antiviral treatment have not been resolved, that is, optimal duration, effect of postpartum therapy, and risk of postpartum alanine aminotransferase (ALT) flare after withdrawal. Will the risk of postpartum hepatitis flares increase after short-term AVT in late pregnancy for maternal HBV infection is discontinued? Is there any correlation between postpartum hepatitis flares and withdrawal time? Will the proportion of postpartum flares be reduced if extending the duration of AVT after delivery? There is an urgent need in this area. This study mainly investigated the safety of antiviral therapy in preventing HBV mother-to-child transmission in pregnant women after discontinuation.

DETAILED DESCRIPTION:
Between June 2015 and December 2017, 111 mothers were enrolled during their visit to the Department of Gynecology and Obstetrics or the Department of Infectious Diseases of the Third Affiliated Hospital of Sun Yat-Sen University in Guangzhou, Guangdong province, China. Pregnant women fulfilling the inclusion and exclusion criteria were offered participation in the study. All pregnant women who opted for AVT need to sign a consent form and started on oral telbivudine (LDT) 600 mg or tenofovir disoproxil fumarate (TDF) 300 mg (as per patients' wishes) daily between gestational weeks 24 and 28. Serum levels of HBV DNA, HBsAg, HBsAb, HBeAg, HBeAb, liver function tests, haematology and renal biochemistry were measured at baseline(i.e. at screening), every 4 weeks after treatment begins, at the time of delivery, and at 1, 2, 3, 6, 12 month postpartum. After delivery, treatment with LDT or TDF was immediately withdrew to the patients with an intention of breastfeeding, while the other patients, without desire of breastfeeding, would subsequently extend antiviral treatment duration to postpartum 6 weeks. All infants were vaccinated with genetically engineered HBV vaccine 20 ug according to a standard vaccination regimen (i.e. within 12h of birth, at week 4 and at week 24) and 200 IU doses of hepatitis B immunoglobulin immediately (within 2h) after birth and at day 15. The infant's HBV serologic status and HBV DNA were tested at birth (before immunization) and again at 7 months. The investigators discussed the postpartum liver function after withdrawal and evaluated the impact of extending the postpartum duration of AVT administered for the prevention of perinatal transmission.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24 and 28 weeks
* Detectable serum HBsAg at the Screening visit and at least 6 months prior
* Serum HBV DNA level >1,000,000 IU/mL at Screening visit
* Alanine aminotransferase (ALT) below the upper limit of normal (ULN; 40 IU/mL)

Exclusion Criteria:

* Patient is co-infected with hepatitis A virus, hepatitis C virus, hepatitis delta virus, hepatitis E virus or HIV.
* Patient has a history of antiviral treatment or concurrent treatment with immunomodulators, cytotoxic drugs, or steroids.
* Patient has clinical signs of threatened miscarriage in early pregnancy.
* Patient has evidence of hepatocellular carcinoma or cirrhosis.
* Patient has evidence of fetal deformity by 3-dimensional ultrasound examination.
* Patient has a husband infected with HBV.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Postpartum flare incidence | From baseline to postpartum 12 months.
  Time-to-event measures. Postpartum flare was defined as an alanine aminotransferase (ALT) rise to three times baseline level or five times ULN (40U/L) within 12 months post-delivery. Maternal would be recorded if postpartum flare occured. At the end of postpartum 12-month follow-up period, postpartum flare incidence was measured.

SECONDARY OUTCOMES:
Time of flare onset | Baseline (i.e. at screening); at the time of delivery; at 1,2,3,6,12 month postpartum.
  Time-to-event measures. Time of the onset of postpartum liver damage.
Proportion of severe flares | Baseline (i.e. at screening); at the time of delivery; at 1,2,3,6,12 month postpartum.
  As per protocol, ALT flares (>5 times baseline level or >10 times ULN) were considered severe adverse events (SAEs).
Peak ALT during flare | Baseline (i.e. at screening); at the time of delivery; at 1,2,3,6,12 month postpartum.
  Peak ALT during postpartum flare.
The rate of perinatal transmission | 7 months after birth.
  Perinatal transmission was established by detectable HBV DNA and HBsAg levels in the peripheral blood of infants at 7 months.
HBV kinetics in patients | Baseline (i.e. at screening); at 4-week intervals after treatment was begun up to delivery; at the time of delivery; at 1,2,3,6,12 month postpartum.
  Changes of HBV viral load in patients treated and not treated with antiviral agents.
The liver function normalization rate | Baseline (i.e. at screening); at 4-week intervals after treatment was begun up to delivery; at the time of delivery; at 1,2,3,6,12 month postpartum.
  Normal liver function was defined as the value of ALT level lower 40U/L.
Maternal HBsAg loss/seroconversion rate | Baseline (i.e. at screening); at 4-week intervals after treatment was begun up to delivery; at the time of delivery; at 1,2,3,6,12 month postpartum.
  Measurement of the proportion of maternal hepatitis B surface antigen loss and seroconversion.
Incidence of perinatal and partum complications | Baseline (i.e. at screening); at 4-week intervals after treatment was begun up to delivery; at the time of delivery; at 1,2,3,6,12 month postpartum.
  Perinatal and partum complications included hypertensive disorders in pregnancy, gestational diabetes mellitus, fetal growth retardation, premature delivery, premature rupture of membrane, and postpartum hemorrhage.
Birth height | At the time of delivery.
  Measurement of infants' height at the time of delivery.
Birth weight | At the time of delivery.
  Measurement of infants' weight at the time of delivery.
Neonate apgar score at 1 minute | At 1 minute after birth.
  Apgar scores of neonates included activity, pulse, grimace, appearance and respiration.
Neonate apgar score at 5 minutes | At 5 minutes after birth.
  Apgar scores of neonates included activity, pulse, grimace, appearance and respiration.
Incidence of deformity | At the time of delivery; at 1, 7, 12 month postpartum.
  The incidence of baby deformity was recorded during the postpartum follow-up period.
Breastfeeding rate | At birth, at 1 and 7 month follow-up.
  Breast feeding status was assessed in all infants during the postpartum follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-liang Gao, PhD, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not available to other researchers.